CLINICAL TRIAL: NCT00002700
Title: A RANDOMIZED PHASE III TRIAL COMPARING DEXAMETHASONE WITH PREDNISONE IN INDUCTION TREATMENT AND BONE MARROW TRANSPLANTATION WITH INTENSIVE MAINTENANCE TREATMENT IN ADOLESCENT AND ADULT ACUTE LYMPHOBLASTIC LEUKEMIA (ALL-4)
Brief Title: Chemotherapy With or Without Bone Marrow Transplantation in Treating Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-06951; EORTC-06951; FRE-LALA-94
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma
Keywords: untreated adult acute lymphoblastic leukemia; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; Mitoxantrone; Prednisolone; Prednisone; Hydrocortisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: leucovorin calcium
Drug: mercaptopurine
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: prednisolone
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells. Bone marrow transplantation can replace immune cells that were destroyed by chemotherapy.

PURPOSE: Randomized phase III trial to study the effectiveness of chemotherapy compared with or without bone marrow transplantation in treating patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the remission induction, toxicity, and duration of remission in patients with newly diagnosed acute lymphoblastic leukemia or lymphoblastic lymphoma treated with prednisone vs dexamethasone plus cyclophosphamide, daunorubicin, and vincristine as induction.
* Compare the survival and disease-free survival of patients treated with autologous bone marrow transplantation (BMT) followed by low- or high-intensity maintenance chemotherapy with cranial irradiation after consolidation.
* Determine the relative and disease-free survival of patients treated with autologous or allogeneic BMT after identical induction, consolidation, and conditioning regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center and risk group (high vs standard).

Induction

* Patients are randomized to 1 of 2 treatment arms.

  * Arm I:Patients receive daunorubicin IV on days 1-3 and 15 and 16; cyclophosphamide (CTX) IV on days 1 and 8; vincristine (VCR) IV on days 1, 8, 15, and 22; and prednisone IV or orally every 8 hours on days 1-7 and 15-21.
  * Arm II: Patients receive daunorubicin, CTX, and VCR as in arm I and dexamethasone IV or orally on days 1-8 and 15-22.
* Patients on both arms without CNS disease at presentation receive CNS prophylaxis comprising methotrexate (MTX) intrathecally (IT) on days 1, 8, 15, and 22. Patients on both arms with CNS disease at presentation receive CNS therapy comprising hydrocortisone (HC) IT and MTX IT alternating with cytarabine (ARA-C) IT twice a week until CSF clears. After induction, patients on both arms proceed to consolidation, regardless of response.

Consolidation

* Patients receive ARA-C IV over 2 hours every 12 hours on days 29-34 and mitoxantrone IV on days 33-35. Patients without CNS disease at presentation receive CNS prophylaxis comprising MTX IT on day 29. Patients with CNS disease at presentation receive CNS therapy comprising HC IT and MTX IT alternating with ARA-C weekly for 6 weeks. Patients who achieve complete response (CR) at day 55-60 receive MTX IV on days 64 and 79, leucovorin calcium IV or orally every 6 hours on days 65-67 and 80-82, and asparaginase IV over 1 hour or intramuscularly on days 65 and 80.
* Standard-risk patients who are under age 20 and achieve CR after day 80 are assigned to arm IV of group A. Patients who achieve CR after day 80 and have a genotypically or phenotypically HLA-matched family donor, a family donor mismatched at only 1 locus (A, B, or DR), or an HLA-matched unrelated donor proceed to group B. Patients who achieve CR after day 80 and are eligible for autologous bone marrow transplantation (BMT) proceed to group A. Patients found to be at extremely high risk are taken off study.

Group A

* Patients are randomized to 1 of 2 treatment arms.

  * Arm III: Autologous bone marrow is harvested. Patients receive bone marrow ablation comprising CTX IV over 1 hour on days -4 and -3 and total body irradiation on day -1. Autologous bone marrow is reinfused on day 0. Beginning at month 8 (4 months after BMT), patients receive first maintenance comprising VCR IV, doxorubicin IV, and dexamethasone IV (VAD) or VCR IV, doxorubicin IV, and prednisolone IV (VAP) on days 1-4 and 29-32. Patients receive second maintenance comprising oral mercaptopurine daily and oral MTX daily beginning at month 10 and continuing through year 3. Patients without CNS disease at presentation receive CNS prophylaxis comprising MTX IT on days 1 and 29. Patients with CNS disease at presentation receive CNS therapy comprising ARA-C IT, MTX IT, and HC IT beginning at 1 month after BMT and continuing monthly for 1 year and then every 3 months through year 3.
  * Arm IV: Patients receive CTX IV and ARA-C IV continuously on day 1, oral mercaptopurine on days 8-28, and oral MTX on days 8, 15, and 22 during months 4, 7, 11, 13, 17, 21, 25, and 29. Patients receive MTX IV over 30 minutes on day 1, leucovorin calcium IV or orally every 6 hours on days 2-4, asparaginase IV over 1 hour or intramuscularly on day 2, oral mercaptopurine on days 8-28, and oral MTX on days 8, 15, and 22 during months 6, 10, 12, 15, 19, 23, and 27. Patients receive VAD or VAP as in arm III beginning at month 8. Patients without CNS disease at presentation receive CNS prophylaxis comprising whole brain radiotherapy and MTX IT on day 1 of radiotherapy during month 5. Patients with CNS disease at presentation receive CNS therapy as in arm III.

Group B

* Allogeneic bone marrow is harvested. Patients receive bone marrow ablation as in arm III beginning on day 100. Allogeneic bone marrow is infused over 15-30 minutes on day 0.

  * Patients in groups A and B with CNS disease at presentation undergo radiotherapy to focal infiltration at entry or concurrently with total body irradiation, or whole brain radiotherapy during maintenance (if no prior CNS irradiation). At any time during the study, patients who develop marrow relapse (more than 5% leukemic blasts in bone marrow on 2 occasions), CNS relapse (blasts in CSF, cranial nerve palsy, or CNS mass), or testis or other extramedullary relapse are taken off study.

PROJECTED ACCRUAL: A total of 392 patients will be accrued for this study within approximately 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia or lymphoblastic lymphoma with more than 30% blasts in bone marrow

PATIENT CHARACTERISTICS:

Age:

* 15 to 60

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin less than 2 mg/dL (unless elevation due to leukemic involvement of liver)

Renal:

* Creatinine less than 2 mg/dL (unless elevation due to leukemic involvement of kidneys)

Cardiovascular:

* No severe cardiac disease

Pulmonary:

* No severe pulmonary disease

Other:

* No severe neurologic or metabolic disease
* HIV negative (if tested)
* No other prior malignancy except nonmelanomatous skin cancer, stage I cervical carcinoma, or other curatively treated malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No prior endocrine therapy

Radiotherapy:

* No prior radiotherapy

Surgery:

* No prior surgery

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 392 (Estimated)
Dates: Start 1995-08; Primary Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roel Willemze, MD, PhD, Study Chair — Leiden University Medical Center; Denis Fiere, MD, Study Chair — Acute Leukemia French Association
Locations (44):
- Belgium (7):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - C.H.U. Saint-Pierre, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Sart-Tilman, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Croatia (2):
  - University Hospital Rebro, Zagreb
  - Medical School/University of Zagreb, Zagreb (Agram)
- University Hospital - Olomouc, Olomouc, Czechia
- France (4):
  - Hopital Edouard Herriot, Lyon
  - Hotel Dieu de Paris, Paris
  - Hopital Necker, Paris
  - Centre Medico-Chirurgical Foch, Suresnes
- Kreiskrankenhaus Meissen, Meissen, Germany
- Italy (21):
  - Ospedale Civile Alessandria, Alessandria
  - Ospedale Civile Avellino, Avellino
  - Universita Degli Studi di Bari Policlinico, Bari
  - A. Perrino Hospital, Brindisi
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Ospedale Santa Croce, Cuneo
  - Policlinico di Careggi, Firenze (Florence)
  - Ospedali Riuniti Foggia, Foggia
  - Ospedale S. Antonio Abate, Gallarate Varese
  - Ospedale Gen. Provinciale Santa Maria Goretti, Latina
  - Ospedale Maggiore Lodi, Lodi
  - Ospedale Di Montefiascone, Montefiascone
  - Ospedale S. Gennaro ASL NA1, Naples (Napoli)
  - Policlinico - Cattedra di Ematologia, Palermo
  - Policlinico Monteluce, Perugia
  - Ospedale San Carlo, Potenza
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Istituto di Ematologia Universita - University di Sassari, Sassari
  - Ospedal SS Annunziata, Taranto
  - Ospedale Molinette, Turin (Torino)
- Netherlands (5):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Maxima Medisch Centrum - locatie Eindhoven, Eindhoven
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
- Hospital Escolar San Joao, Porto, Portugal
- Institute of Hematology & Transfusiology, University Hospital, Bratislava, Slovakia
- Ibn-i Sina Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Reman O, Pigneux A, Huguet F, Vey N, Delannoy A, Fegueux N, de Botton S, Stamatoullas A, Tournilhac O, Buzyn A, Charrin C, Boucheix C, Gabert J, Lheritier V, Vernant JP, Fiere D, Dombret H, Thomas X; GET-LALA group. Central nervous system involvement in adult acute lymphoblastic leukemia at diagnosis and/or at first relapse: results from the GET-LALA group. Leuk Res. 2008 Nov;32(11):1741-50. doi: 10.1016/j.leukres.2008.04.011. Epub 2008 May 27. PMID 18508120
- [Background] Tavernier E, Le QH, de Botton S, Dhedin N, Bulabois CE, Reman O, Vey N, Lheritier V, Dombret H, Thomas X. Secondary or concomitant neoplasms among adults diagnosed with acute lymphoblastic leukemia and treated according to the LALA-87 and LALA-94 trials. Cancer. 2007 Dec 15;110(12):2747-55. doi: 10.1002/cncr.23097. PMID 17963265
- [Background] Dhedin N, Dombret H, Thomas X, Lheritier V, Boiron JM, Rigal-Huguet F, Vey N, Kuentz M, Reman O, Witz F, Delannoy A, Kovacsovics T, Bradstock K, Charrin C, Boucheix C, Gabert J, Blaise D, Fiere D, Vernant JP. Autologous stem cell transplantation in adults with acute lymphoblastic leukemia in first complete remission: analysis of the LALA-85, -87 and -94 trials. Leukemia. 2006 Feb;20(2):336-44. doi: 10.1038/sj.leu.2404065. PMID 16357838
- [Background] Picard C, Hayette S, Bilhou-Nabera C, Cayuela JM, Delabesse E, Frenoy N, Preudhomme C, Dupont M, Bastard C, Bories D, Vaerman JL, Davi F, Dastugue N, Raynaud S, Lafage M, Deschaseaux F, Fest T, Gaub MP, Lheritier V, Thomas X, Charrin C, Boucheix C, Dombret H, Macintyre E, Fiere D, Gabert J. Prospective multicentric molecular study for poor prognosis fusion transcripts at diagnosis in adult B-lineage ALL patients: the LALA 94 experience. Leukemia. 2006 Dec;20(12):2178-81. doi: 10.1038/sj.leu.2404408. Epub 2006 Oct 12. No abstract available. PMID 17039237
- [Background] Charrin C, Thomas X, Ffrench M, Le QH, Andrieux J, Mozziconacci MJ, Lai JL, Bilhou-Nabera C, Michaux L, Bernheim A, Bastard C, Mossafa H, Perot C, Maarek O, Boucheix C, Lheritier V, Delannoy A, Fiere D, Dastugue N. A report from the LALA-94 and LALA-SA groups on hypodiploidy with 30 to 39 chromosomes and near-triploidy: 2 possible expressions of a sole entity conferring poor prognosis in adult acute lymphoblastic leukemia (ALL). Blood. 2004 Oct 15;104(8):2444-51. doi: 10.1182/blood-2003-04-1299. Epub 2004 Mar 23. PMID 15039281
- [Background] Boissel N, Auclerc MF, Lheritier V, Perel Y, Thomas X, Leblanc T, Rousselot P, Cayuela JM, Gabert J, Fegueux N, Piguet C, Huguet-Rigal F, Berthou C, Boiron JM, Pautas C, Michel G, Fiere D, Leverger G, Dombret H, Baruchel A. Should adolescents with acute lymphoblastic leukemia be treated as old children or young adults? Comparison of the French FRALLE-93 and LALA-94 trials. J Clin Oncol. 2003 Mar 1;21(5):774-80. doi: 10.1200/JCO.2003.02.053. Epub 2003 Mar 1. PMID 12610173
- [Result] Labar B, Suciu S, Willemze R, Muus P, Marie JP, Fillet G, Berneman Z, Jaksic B, Feremans W, Bron D, Sinnige H, Mistrik M, Vreugdenhil G, De Bock R, Nemet D, Gilotay C, Amadori S, de Witte T; EORTC Leukemia Group. Dexamethasone compared to prednisolone for adults with acute lymphoblastic leukemia or lymphoblastic lymphoma: final results of the ALL-4 randomized, phase III trial of the EORTC Leukemia Group. Haematologica. 2010 Sep;95(9):1489-95. doi: 10.3324/haematol.2009.018580. Epub 2010 Apr 7. PMID 20378563
- [Result] Le QH, Thomas X, Ecochard R, Iwaz J, Lheritier V, Michallet M, Fiere D. Proportion of long-term event-free survivors and lifetime of adult patients not cured after a standard acute lymphoblastic leukemia therapeutic program: adult acute lymphoblastic leukemia-94 trial. Cancer. 2007 May 15;109(10):2058-67. doi: 10.1002/cncr.22632. PMID 17407135
- [Result] Tavernier E, Boiron JM, Huguet F, Bradstock K, Vey N, Kovacsovics T, Delannoy A, Fegueux N, Fenaux P, Stamatoullas A, Tournilhac O, Buzyn A, Reman O, Charrin C, Boucheix C, Gabert J, Lheritier V, Vernant JP, Dombret H, Thomas X; GET-LALA Group; Swiss Group for Clinical Cancer Research SAKK; Australasian Leukaemia and Lymphoma Group. Outcome of treatment after first relapse in adults with acute lymphoblastic leukemia initially treated by the LALA-94 trial. Leukemia. 2007 Sep;21(9):1907-14. doi: 10.1038/sj.leu.2404824. Epub 2007 Jul 5. PMID 17611565
- [Result] Vey N, Thomas X, Picard C, Kovascovicz T, Charin C, Cayuela JM, Dombret H, Dastugue N, Huguet F, Bastard C, Stamatoulas A, Giollant M, Tournilhac O, Macintyre E, Buzyn A, Bories D, Kuentz M, Dreyfus F, Delannoy A, Raynaud S, Gratecos N, Bordessoule D, de Botton S, Preudhomme C, Reman O, Troussard X, Pigneux A, Bilhou C, Vernant JP, Boucheix C, Gabert J; GET-LALA Group the Swiss Group for Clinical Cancer Research (SAKK). Allogeneic stem cell transplantation improves the outcome of adults with t(1;19)/E2A-PBX1 and t(4;11)/MLL-AF4 positive B-cell acute lymphoblastic leukemia: results of the prospective multicenter LALA-94 study. Leukemia. 2006 Dec;20(12):2155-61. doi: 10.1038/sj.leu.2404420. Epub 2006 Oct 12. PMID 17039234
- [Result] Asnafi V, Buzyn A, Thomas X, Huguet F, Vey N, Boiron JM, Reman O, Cayuela JM, Lheritier V, Vernant JP, Fiere D, Macintyre E, Dombret H. Impact of TCR status and genotype on outcome in adult T-cell acute lymphoblastic leukemia: a LALA-94 study. Blood. 2005 Apr 15;105(8):3072-8. doi: 10.1182/blood-2004-09-3666. Epub 2005 Jan 6. PMID 15637138
- [Result] Thomas X, Boiron JM, Huguet F, Dombret H, Bradstock K, Vey N, Kovacsovics T, Delannoy A, Fegueux N, Fenaux P, Stamatoullas A, Vernant JP, Tournilhac O, Buzyn A, Reman O, Charrin C, Boucheix C, Gabert J, Lheritier V, Fiere D. Outcome of treatment in adults with acute lymphoblastic leukemia: analysis of the LALA-94 trial. J Clin Oncol. 2004 Oct 15;22(20):4075-86. doi: 10.1200/JCO.2004.10.050. Epub 2004 Sep 7. PMID 15353542
- [Result] Asnafi V, Buzyn A, Thomas X, et al.: Impact of immunophenotype and genotype on outcome in LALA94 T-ALLs: toward risk adapted stratification of adult T-ALL. [Abstract] Blood 102 (11): A-67, 2003.
- [Result] Dombret H, Gabert J, Boiron JM, Rigal-Huguet F, Blaise D, Thomas X, Delannoy A, Buzyn A, Bilhou-Nabera C, Cayuela JM, Fenaux P, Bourhis JH, Fegueux N, Charrin C, Boucheix C, Lheritier V, Esperou H, MacIntyre E, Vernant JP, Fiere D; Groupe d'Etude et de Traitement de la Leucemie Aigue Lymphoblastique de l'Adulte (GET-LALA Group). Outcome of treatment in adults with Philadelphia chromosome-positive acute lymphoblastic leukemia--results of the prospective multicenter LALA-94 trial. Blood. 2002 Oct 1;100(7):2357-66. doi: 10.1182/blood-2002-03-0704. PMID 12239143